CLINICAL TRIAL: NCT07199023
Title: Dietary Restriction Efficiency Assessment of Different Hypoallergenic Formulas in Patients With Suspected Cow's Milk Protein Allergy
Brief Title: Dietary Restriction Efficiency Assessment in CMPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Collaborators: Guangzhou Women and Children's Medical Center (Other); Beijing Children's Hospital (Other); Peking University Third Hospital (Other); Guangdong Provincial People's Hospital (Other); Chengdu Women's and Children's Central Hospital (Other); Guiyang Maternity and Child Health Care Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DREAM-CHINA
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-08

CONDITIONS: Cow's Milk Protein Allergy
Keywords: Amino Acid Formula; Extended Hydrolyzed Formula; Cow's milk protein allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either an amino acid formula (AAF) or an extensively hydrolyzed formula (eHF) during the diagnostic elimination diet phase. Both groups will follow at least 2 weeks of formula-based feeding. Infants in the eHF group who do not show symptom improvement may switch to AAF for another 2 weeks. Symptom improvement will be evaluated to determine eligibility for an oral food challenge (OFC) to confirm the diagnosis of cow's milk protein allergy (CMPA).
Masking Description: Masking Description
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amino Acid Formula Group (AAF Group) (Active Comparator): Participants in this group will receive an amino acid-based formula (AAF) for at least 2 weeks during the elimination diet phase. If symptoms improve, participants will undergo an oral food challenge (OFC) to confirm the diagnosis of cow's milk protein allergy (CMPA). If symptoms do not improve after 4 weeks, CMPA will be ruled out.
  Interventions: Dietary Supplement: Amino Acid Formula (AAF)
- Extensively Hydrolyzed Formula Group (eHF Group) (Experimental): Participants in this group will receive an extensively hydrolyzed formula (eHF) for at least 2 weeks during the elimination diet phase. If symptoms improve, OFC will be conducted to confirm CMPA diagnosis. If no improvement is observed, participants may switch to AAF for another 2 weeks of intervention.
  Interventions: Dietary Supplement: Extensively Hydrolyzed Formula (eHF)

INTERVENTIONS:
Dietary Supplement: Amino Acid Formula (AAF) — A formula composed of 100% free amino acids with no intact cow's milk protein. Participants will be fed AAF ad libitum according to their nutritional needs. Daily intake and symptoms will be recorded through an electronic diary (eCOA).
  Arms: Amino Acid Formula Group (AAF Group)
Dietary Supplement: Extensively Hydrolyzed Formula (eHF) — A formula in which cow's milk proteins are broken down into small peptides through enzymatic hydrolysis, reducing allergenicity. Participants will be fed eHF ad libitum based on their nutritional needs. Intake and symptoms will be tracked through an electronic diary (eCOA).
  Arms: Extensively Hydrolyzed Formula Group (eHF Group)

SUMMARY:
This clinical trial aims to evaluate and compare the efficacy of amino acid formula (AAF) and extensively hydrolyzed formula (eHF) in relieving symptoms in infants suspected of cow's milk protein allergy (CMPA) during the diagnostic elimination diet phase. The study will also assess treatment compliance, economic costs, and develop a CMPA screening score suitable for Chinese infants.

Eligible infants (0-6 months old) will be randomized to receive either AAF or eHF for at least 2 weeks. Symptom improvement will be evaluated, followed by an oral food challenge (OFC) to confirm CMPA diagnosis. Infants in the eHF group who do not improve may switch to AAF for further evaluation. The total duration of participation is approximately 6 to 8 weeks.

The study aims to provide evidence-based data to optimize diagnostic pathways and improve quality of life for infants with CMPA.

DETAILED DESCRIPTION:
Cow's milk protein allergy (CMPA) is one of the most common food allergies in infants, with a prevalence of approximately 2.5-3.0% globally and 0.83-3.5% in China. Accurate diagnosis is often challenging due to the non-specific and variable symptoms, which may involve gastrointestinal, dermatologic, or respiratory systems. The current diagnostic gold standard involves an elimination diet followed by an oral food challenge (OFC). However, the choice of formula during the elimination phase may affect both symptom relief and diagnostic accuracy.

This multicenter, randomized, open-label controlled trial (DREAM-CHINA) is designed to evaluate the clinical efficacy of two hypoallergenic formulas-amino acid formula (AAF) and extensively hydrolyzed formula (eHF)-in the diagnostic elimination diet phase for infants suspected of having CMPA. The study also aims to compare the two formulas in terms of symptom improvement rate, economic burden, treatment compliance, and formula acceptance.

A total of 320 infants aged 0-6 months with suspected CMPA will be enrolled and randomized (1:1) to receive either AAF or eHF for at least 2 weeks. Infants whose symptoms significantly improve will undergo an OFC to confirm the diagnosis. Those in the eHF group who do not show improvement may switch to AAF for an additional 2 weeks before undergoing OFC.

Record the speed of symptom improvement after eliminating the diet, and evaluate the diagnosis rate of CMPA through OFC, the time of symptom improvement, safety results, and the effectiveness of symptom-based screening tools for CMPA in Chinese infants.

Throughout the study, data will be collected via electronic diaries (eCOA), clinical assessments, and standardized symptom scoring tools (e.g., CoMiSS). Regular follow-ups will monitor anthropometric growth, symptom progression, and adverse events. This study seeks to provide high-quality evidence for optimizing clinical decision-making and improving the diagnostic process for CMPA in Chinese infants.

ELIGIBILITY:
Inclusion Criteria:

Infants aged 0-6 months; Diagnosed with suspected CMPA at the time of presentation; Artificially or mixed-feeding; Parents willing to sign a written informed consent and comply with the study protocol.

Exclusion Criteria:

Infants currently receiving eHF or AAF formula; Mixed-feeding infants whose current daily formula intake is less than 50% of their total milk intake or less than 200 ml; Infants who have already started adding complementary foods; Infants who have experienced severe food allergy symptoms such as shock, severe vomiting, etc. after taking cow's milk protein; Infants with clinical manifestations of systemic allergic reaction or respiratory difficulties such as acute laryngeal edema or bronchial obstruction; Infants who have used prednisolone or anti-allergic drugs in the past 2 weeks; Infants with contraindications to eHF or AAF formula; Infants whose parents are unable to fully report the occurrence of possible symptoms (e.g., insufficient language skills); Infants with other serious diseases, including but not limited to growth retardation, metabolic disorders, kidney disease, congenital heart disease, medical conditions requiring hospitalization for more than 2 weeks, etc.; Infants whose mothers are unable to avoid necessary foods when mixed-feeding.

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients with significantly improved symptoms after EDA in the two groups | 2 weeks after enrolled
  The criteria for improvement are:
  * A ≥50% reduction in the Diarrhea and Blood Stool Score. ② A ≥50% reduction in the CoMiSS Score. ③ Marked improvement or resolution of original gastrointestinal and skin symptoms, such as spit-up, vomiting, diarrhea, abdominal distension, abdominal pain, and reflux.

SECONDARY OUTCOMES:
The number of days it takes for the child to achieve significant improvement in symptoms | 2 weeks after enrolled
  The number of days from the start of the intervention until the child first meets the aforementioned 'marked symptom improvement' criteria.

OTHER OUTCOMES:
CMPA diagnosis rate (OFC positive rate) | 2 weeks after enrolled
  The proportion of cases with positive EDA results and positive OFC
Sensitivity and validity of CMPA score | 2 weeks after enrolled
  Compare the diagnostic performance of the CMPA scores in OFC-positive and OFC-negative groups.

CONTACTS AND LOCATIONS:
Overall Officials: Chundi Xu, Principal Investigator — Ruijin Hospital